CLINICAL TRIAL: NCT01573351
Title: A Phase 3, Open-Label Study With Asunaprevir and Daclatasvir Plus Peginterferon Alfa-2a (Pegasys) and Ribavirin (Copegus) (P/R) (QUAD) for Subjects Who Are Null or Partial Responders to Peginterferon Alfa 2a or 2b Plus Ribavirin With Chronic Hepatitis C Genotypes 1 or 4 Infection
Brief Title: Phase III Hallmark QUAD: ASV+DCV+Peg+Rib (Nulls/Partials)
Acronym: Hallmark QUAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI447-029; 2011-005422-21 (EudraCT Number)
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — asunaprevir; daclatasvir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- QUAD: Asunaprevir+Daclatasvir+Peg-interferon Alfa-2a+Ribavirin (Experimental): Asunaprevir: Capsule, Oral, 100 mg, Twice daily, 24 weeks
  Daclatasvir: Tablet, Oral, 60 mg, Once daily, 24 weeks
  Peg-interferon Alfa-2a: Injection, subcutaneous (SC), 180 mcg/0.5 mL, Once weekly, 24 weeks
  Ribavirin: Tablet, Oral, 1000 mg/1200 mg (total daily dose), 24 weeks
  Interventions: Drug: Asunaprevir; Drug: Daclatasvir; Drug: Peg-interferon Alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Asunaprevir
  Other Names: BMS-650032
Drug: Daclatasvir
  Other Names: BMS-790052
Drug: Peg-interferon Alfa-2a
  Other Names: Pegasys®
Drug: Ribavirin
  Other Names: Copegus®

SUMMARY:
The purpose of this study is to assess efficacy, as determined by the proportion of subjects with Sustained Virologic Response at Post-Treatment Week 12 (SVR12), defined as Hepatitis C virus (HCV) Ribonucleic acid (RNA) < Limit of quantitation (LOQ) at post-treatment Week 12.

DETAILED DESCRIPTION:
* ASV = Asunaprevir (BMS-650032)
* DCV = Daclatasvir (BMS-790052)
* Peg = Peg-interferon Alfa-2a (PegIFN)
* Rib = Ribavirin (RBV)

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥ 18 years of age
* HCV Genotype 1 or 4 who previously failed treatment with Peginterferon alfa-2a or peginterferon alfa-2b and Ribavirin (P/R), classified as previous null and partial responders based on previous therapy
* HCV RNA ≥ 10,000 IU/mL
* Seronegative for Human immunodeficiency virus (HIV) and Hepatitis B surface antigen (HBsAg)
* Subjects with compensated cirrhosis are permitted (compensated cirrhotics are capped at approximately 25% of treated population)

Exclusion Criteria:

* Prior treatment of HCV with HCV direct acting antiviral (DAA)
* Evidence of a medical condition contributing to chronic liver disease other than HCV
* Evidence of decompensated liver disease including, but not limited to, a history or presence of ascites, bleeding varices, or hepatic encephalopathy
* Diagnosed or suspected hepatocellular carcinoma or other malignancies
* Uncontrolled diabetes or hypertension
* Total bilirubin ≥ 34 μmol/L (or ≥ 2 mg/dL) unless subject has a documented history of Gilbert's disease
* Alanine aminotransferase (ALT) ≥ 5x Upper limit of normal (ULN)
* Albumin < 3.5 g/dL (35 g/L)
* Alpha Fetoprotein (AFP) > 100 ng/mL (>82.6 IU/mL) or ≥ 50 and ≤ 100 ng/mL requires a liver ultrasound and subjects with findings suspicious of Hepatocellular carcinoma (HCC) are excluded
* Absolute neutrophil count (ANC) < 1.5 x 1000,000,000 cells/L (< 1.2 x 1000,000,000 cells/L for Black/African-Americans)
* Platelets < 90 x 1000,000,000 cells/L
* Hemoglobin < 12 g/dL for females or < 13 g/dL for males
* Any criteria that would exclude the subject from receiving P/R

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Proportion of genotype 1 subjects with SVR12, defined as HCV RNA < LOQ at post-treatment Week 12, for all subjects infected with HCV genotype 1 | At 12 weeks post-treatment

SECONDARY OUTCOMES:
On-treatment safety, as measured by frequency of Serious Adverse Events (SAEs) and discontinuations due to Adverse Events (AEs) through the end of treatment | Through the end of treatment (maximum up to 24 weeks) plus 7 days
Proportion of subjects with SVR12 (HCV RNA < LOQ at post-treatment Week 12) by the rs12979860 single nucleotide polymorphisms (SNP) in the IL28 gene | At post-treatment Week 12
Proportion of subjects with HCV RNA undetectable | Weeks 1, 2, 4, 6, 8 and 12; at both Weeks 4 and 12 [Extended rapid virologic response (eRVR)], end of treatment (up to 24 weeks), post-treatment Week 12 or post-treatment Week 24
Proportion of subjects with HCV RNA < LOQ | Weeks 1, 2, 4, 6, 8 and 12; at both Weeks 4 and 12, end of treatment (up to 24 weeks), post-treatment Week 24 (SVR24)
Proportion of patients with SVR12 (HCV RNA < LOQ at post-treatment Week 12) for HCV genotype 4 subjects | Post-treatment Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (73):
- United States (20):
  - Alabama Liver & Digestive Specialists (Alds), Montgomery, Alabama
  - Scripps Clinic, La Jolla, California
  - Scpmg/ Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - University Of Colorado Denver And Hospital, Aurora, Colorado
  - South Denver Gastroenterology, Pc, Englewood, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - University Of Miami Schiff Center For Liver Diseases, Miami, Florida
  - University Of Chicago Medical Center, Chicago, Illinois
  - North Shore University Hospital, Manhasset, New York
  - University Of North Carolina At Chapel Hill School Of Med, Chapel Hill, North Carolina
  - University Of Cincinnati, Cincinnati, Ohio
  - Options Health Research, Llc, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Gastro One, Germantown, Tennessee
  - Baylor College Of Medicine, Houston, Texas
  - Texas Liver Institute, San Antonio, Texas
  - Mcguire Dvamc, Richmond, Virginia
  - Dean Clinic, Madison, Wisconsin
- Argentina (3):
  - Local Institution, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, Prov. Buenos Aires, Buenos Aires
- Canada (5):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
- Denmark (3):
  - Local Institution, Aalborg
  - Local Institution, Hvidovre
  - Local Institution, Odense
- France (5):
  - Local Institution, Créteil
  - Local Institution, Montpellier
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Pessac
- Germany (7):
  - Local Institution, Berlin
  - Local Institution, Düsseldorf
  - Local Institution, Frankfurt
  - Local Institution, Freiburg im Breisgau
  - Local Institution, Hamburg
  - Local Institution, Heidelberg
  - Local Institution, Tübingen
- Italy (4):
  - Local Institution, Brescia
  - Local Institution, Cisanello (pisa)
  - Local Institution, Milan
  - Local Institution, Palermo
- Mexico (2):
  - Local Institution, Mexico City, Mexico City
  - Local Institution, México, State of Mexico
- Netherlands (2):
  - Local Institution, Amsterdam
  - Local Institution, Rotterdam
- Russia (4):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Stavropol
  - Local Institution, Tyumen
- South Korea (6):
  - Local Institution, Bucheon-si
  - Local Institution, Busan
  - Local Institution, Daegu
  - Local Institution, Gyeongsangnam-do
  - Local Institution, Incheon
  - Local Institution, Seoul
- Spain (4):
  - Local Institution, Alcorcón
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Seville
- Sweden (2):
  - Local Institution, Gvteborg
  - Local Institution, Stockholm
- Switzerland (2):
  - Local Institution, Bern
  - Local Institution, Lausanne
- Taiwan (4):
  - Local Institution, Chiayi City
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
  - Local Institution, Taipei

REFERENCES:
- [Derived] Jensen D, Sherman KE, Hezode C, Pol S, Zeuzem S, de Ledinghen V, Tran A, Elkhashab M, Younes ZH, Kugelmas M, Mauss S, Everson G, Luketic V, Vierling J, Serfaty L, Brunetto M, Heo J, Bernstein D, McPhee F, Hennicken D, Mendez P, Hughes E, Noviello S; HALLMARK-QUAD Study Team. Daclatasvir and asunaprevir plus peginterferon alfa and ribavirin in HCV genotype 1 or 4 non-responders. J Hepatol. 2015 Jul;63(1):30-7. doi: 10.1016/j.jhep.2015.02.018. Epub 2015 Feb 19. PMID 25703086
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx